CLINICAL TRIAL: NCT03439202
Title: The Effects of Low Intensity Exercise in Hypobaric vs. Normobaric Normoxic and Hypoxic Conditions on Baroreflex Sensitivity, Physiological Responses and Cerebral Functions in Pilots.
Brief Title: Low Intensity Exercise in Different Normobaric/Hypobaric Normoxic/Hypoxic Conditions.
Acronym: Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fliegerärztliches Institut (Other)
Collaborators: University of Lausanne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-00006
Record Dates: First submitted 2018-01-26; First posted 2018-02-20 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Baro-reflex Sensitivity; Heart Rate Variability; EEG, Microstates; Cerebral Blood Flow Regulation; Cerebral Oxygenation; Oxygen Saturation; Concentration Performance
Keywords: Hypoxia; Baro-reflex sensitivity; Low-intensity exercise; Hear rate variability; EEG; Concentration performance
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: Crossover randomized study
Masking Description: No drug and no arm are used for this study. This is a clinical study, because subjects are exposed to hypoxic conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- No arm used (Other): No drug use for this study. No arm used in this study. Subjects are exposed to hypoxic conditions (clinical study).
  Interventions: Other: Hypoxia

INTERVENTIONS:
Other: Hypoxia — Subject will conduct low-intensity exercise on a bike in different hypoxic conditions.
  Other Names: Low-intensity cycling exercise

SUMMARY:
The main goal of this project is to investigate how low intensity cycling exercise (1.5W/kg, for 6 minutes) influences cerebral functions, such as: Cerebral blood flow, oxygenation, and other physiological variables in different normobaric and hypobaric hypoxic conditions.

DETAILED DESCRIPTION:
Subjects will bike at 1W/kg for 6 minutes at different simulated altitude level in the hypobaric chamber at the FAI in Dübendorf. Concentration performance also will be measured to better understand how hypobaric and hypoxia conditions may affect physiological responses, cerebral and cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* Study Indication
* Male and Female subjects from 18 years to 40 years of age
* Healthy volunteer
* Signed Informed Consent after being informed

Exclusion Criteria:

* Contraindications to the study intervention.
* Define drugs, treatments or interventions not allowed during the study or for specific periods of time prior to the intervention,
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Known or suspected non-compliance, drug or alcohol abuse,
* Previous problem with hypoxia or altitude exposure,
* Known pathologies/diseases
* Relevant medical disorders
* Anemia or poor health
* History of flight sickness

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Baro-reflex sensitivity | 6 minutes per record.
  To test the strength of relationship between RR interval and systolic blood pressure in human. Measurement before and after low intensity exercise in each condition.

SECONDARY OUTCOMES:
Concentration performance | 4 minutes per test
  Subjects will conduct a concentration test in each condition.
EEG microstates | 6 minutes per record
  Microstates analysis to investigate how electrical cerebral activity is affected at rest in hypoxia and influenced by low intensity cycling exercise.
Heart rate variability (HRV) | 6 minutes per record
  To investigate about stress (sympathetic and parasympathetic activation) in each condition tested.
Cerebral blood flow | 6 minutes per record.
  Regulation of cerebral blood flow in hypoxia at rest and during low-intensity exercise. Measurement before, during and after low intensity exercise in each condition. 6 minutes recording per measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Bron, Dr. med., Principal Investigator — Aeromedical Center
Locations (1):
- Aeromedical Center / Fliegerärztliches Institut, Dübendorf, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No